CLINICAL TRIAL: NCT01382147
Title: A Randomized, Risk and Age Adapted Comparison of the Dose-Dense Regimen S-HAM (Sequential High Dose Cytosine Arabinoside and Mitoxantrone) Versus Standard Double Induction for Initial Chemotherapy of Adult Patients With Acute Myeloid Leukemia
Brief Title: Evaluation of "Dose-dense Therapy" by S-HAM in Comparison to Conventionally Timed Double Induction in Patients With Acute Myeloid Leukemia (AML)
Acronym: AMLCG 2008
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Dr. Wolfgang Hiddemann (Other)
Collaborators: Kompetenznetz Leukämien (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. Wolfgang Hiddemann, Director of the Department of Medicine III, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-003103-12
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Mitoxantrone; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-HAM (Experimental): S-HAM (S-HAMescalated for younger patients and S-HAMbasis for elderly patients)
  Interventions: Drug: Ara-C, Mitoxantrone, Daunorubicin, Thioguanin
- TAD-HAM (younger) or HAM-HAM (elderly) (Active Comparator): is TAD-9 - HAM for younger patients (with 2 mandatory induction cycles) and HAM (- HAM) for the elderly patients with the second HAM cycle only applied in the case of inadequate blast clearance (> 5%) in the day 16 bone marrow aspirate
  Interventions: Drug: Ara-C, Mitoxantrone, Daunorubicin, Thioguanin

INTERVENTIONS:
Drug: Ara-C, Mitoxantrone, Daunorubicin, Thioguanin — Chemotherapy

SUMMARY:
Evaluation weather early chemotherapy attempts for remission induction can improve the results of patients with Acute Myeloid Leukemia (AML), as compared to the standard group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML (except acute promyelocytic leukemia) according to the WHO classification including patients with secondary AML and AML after preceding hematologic disorders
* Age 18 years or older
* Informed consent. Before any study specific procedure including randomisation is done or before study medication is administered, the subject, or legally acceptable representative, must have given written informed consent for participation in the study.

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)
* Previous or concurrent malignancies other than AML
* Previous treatment with colony-stimulating factors, interleukins or interferons
* Known hypersensitivity to Escherichia coli derived products (e.g. Filgrastim, HUMULIN® Insulin, L-Asparaginase, HUMATROPE® Growth Hormone, INTRON A®)
* Antibody-based or cell-based immunotherapies
* Respiratory insufficiency with pO2 <60 mmHg
* Heart failure NYHA III° or IV°
* Elevated creatinine >2.0 mg/dl
* Elevated bilirubin >2.0 mg/dl
* Pregnancy or lactation
* Females without adequate contraception
* Known HIV and/or hepatitis C infection
* Severe neurologic or psychiatric disease
* Psychiatric, addictive, or any disorder, which compromises ability to give truly informed consent for participation in this study
* Concerns for subject's compliance with the protocol procedures
* Lack of willingness to record and circulate personal disease-related informations defined in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate, aiming at a 15% increase in the CR/PR rate by S-HAM induction versus conventional double induction [TAD - HAM for younger patients, HAM (- HAM) for elderly patients]. | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hiddemann, Prof. Dr., Principal Investigator — Hospital of the University of Munich
Locations (32):
- Germany (32):
  - Vinzenz-Pallotti-Hospital, Innere Abteilung, Bergisch Gladbach
  - St. Hedwig Krankenhaus, Abteilung Innere Medizin, Berlin
  - Vivantes Klinikum Neukoelln, Innere Medizin - Haematologie und Onkologie, Berlin
  - HELIOS Klinikum Berlin-Buch, Klinik für Haematologie, Onkologie und Tumorimmunologie, Berlin
  - Vivantes Klinikum Spandau, Klinik fuer Innere Medizin, Haematologie, Onkologie, Gastroenterologie und Palliativmedizin, Berlin
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Evangelisches Krankenhaus Bielefeld gGmbH, Klinik fuer Innere Medizin, Haematologie, Onkologie und Palliativmedizin, Bielefeld
  - Augusta-Krankenanstalt, Klinik fuer Haematologie, Onkologie und Palliativmedizin, Bochum
  - Evangelische Kliniken Bonn gGmbH, Johanniter Krankenhaus, Innere Medizin I, Bonn
  - Knappschaftskrankenhaus Bottrop, Klinik fuer Innere Medizin, Bottrop
  - Universitaetsklinikum Köln, Klinik I fuer Innere Medizin, Cologne
  - St.-Johannes Hospital Dortmund, Klinik fuer Innere Medizin II, Dortmund
  - St.-Antonius-Hospital Eschweiler, Klinik fuer Haematologie und internistische Onkologie, Eschweiler
  - Klinikum Frankfurt / Oder GmbH, Medizinische Klinik I, Frankfurt (Oder)
  - St.-Josef-Hospital Gelsenkirchen-Horst, Klinik für Medizinische und Radiologische Onkologie, Hämatologie und Palliativmedizin, Gelsenkirchen
  - Städtisches Klinikum Gütersloh, Medizinische Klinik II, Gütersloh
  - Kath. Krankenhaus Hagen GmbH, Klinik fuer Haematologie und Onkologie, Hagen
  - Klinikum Herford, Medizinische Klinik II, Herford
  - Klinikum Idar-Oberstein GmbH, Innere Medizin I, Abteilung Haematologie / Onkologie, Îdar-Oberstein
  - Klinikum Leverkusen gGmbH, Medizinische Klinik III, Leverkusen
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Medizinische Klinik A, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Medizinische Klinik I, Haematologie / Onkologie, Luebbeck
  - Medizinische Fakultaet Mannheim der Universitaet Heidelberg, III. Medizinische Klinik Haematologie und Internistische Onkologie, Mannheim
  - Carl-von-Basedow-Klinikum Saalekreis GmbH, Medizinische Klinik II, Merseburg
  - Krankenhaus Maria Hilf GmbH, Krankenhaus St. Franziskus, Medizinische Klinik I, Mönchengladbach
  - Klinikum der Universitaet Muenchen Medizinische Klinik und Polikklinik III, München
  - Staedtisches Klinikum Harlaching, Klinik für Onkologie und Haematologie, München
  - Klinikum Osnabrück, Klinik fuer Haematologie / Onkologie, Osnabrück
  - Brüderkrankenhaus St. Josef Paderborn, Klinik fuer Haematologie / Onkologie, Paderborn
  - Krankenhaus Barmherzige Brüder , Klinik fuer internistische Onkologie und Haematologie, Regensburg
  - St.-Marien-Krankenhaus Siegen gem. GmbH, Medizinische Klinik III, Siegen
  - Stiftung Deutsche Klinik für Diagnostik GmbH, Zentrum fuer Knochenmark- und Stammzelltransplantation, Wiesbaden

REFERENCES:
- [Derived] Archer KJ, Fu H, Mrozek K, Nicolet D, Mims AS, Uy GL, Stock W, Byrd JC, Hiddemann W, Braess J, Spiekermann K, Metzeler KH, Herold T, Eisfeld AK. Identifying long-term survivors and those at higher or lower risk of relapse among patients with cytogenetically normal acute myeloid leukemia using a high-dimensional mixture cure model. J Hematol Oncol. 2024 May 3;17(1):28. doi: 10.1186/s13045-024-01553-6. PMID 38702786
- [Derived] Pastore F, Gittinger H, Raab S, Tschuri S, Ksienzyk B, Konstandin NP, Schneider S, Rothenberg-Thurley M, Horny HP, Werner M, Sauerland MC, Amler S, Gorlich D, Berdel WE, Wormann B, Braess J, Hiddemann W, Tischer J, Herold T, Metzeler KH, Spiekermann K. Acute megakaryoblastic leukaemia shows high frequency of chromosome 1q aberrations and dismal outcome. Br J Haematol. 2023 Sep;202(6):1165-1177. doi: 10.1111/bjh.18982. Epub 2023 Jul 16. PMID 37455345
- [Derived] Kunadt D, Stasik S, Metzeler KH, Rollig C, Schliemann C, Greif PA, Spiekermann K, Rothenberg-Thurley M, Krug U, Braess J, Kramer A, Hochhaus A, Scholl S, Hilgendorf I, Brummendorf TH, Jost E, Steffen B, Bug G, Einsele H, Gorlich D, Sauerland C, Schafer-Eckart K, Krause SW, Hanel M, Hanoun M, Kaufmann M, Wormann B, Kramer M, Sockel K, Egger-Heidrich K, Herold T, Ehninger G, Burchert A, Platzbecker U, Berdel WE, Muller-Tidow C, Hiddemann W, Serve H, Stelljes M, Baldus CD, Neubauer A, Schetelig J, Thiede C, Bornhauser M, Middeke JM, Stolzel F; A. M. L. Cooperative Group (AMLCG), Study Alliance Leukemia (SAL). Impact of IDH1 and IDH2 mutational subgroups in AML patients after allogeneic stem cell transplantation. J Hematol Oncol. 2022 Sep 5;15(1):126. doi: 10.1186/s13045-022-01339-8. PMID 36064577
- [Derived] Konstandin NP, Pastore F, Herold T, Dufour A, Rothenberg-Thurley M, Hinrichsen T, Ksienzyk B, Tschuri S, Schneider S, Hoster E, Berdel WE, Woermann BJ, Sauerland MC, Braess J, Bohlander SK, Klein HG, Hiddemann W, Metzeler KH, Spiekermann K. Genetic heterogeneity of cytogenetically normal AML with mutations of CEBPA. Blood Adv. 2018 Oct 23;2(20):2724-2731. doi: 10.1182/bloodadvances.2018016840. PMID 30337300
- [Derived] Hubmann M, Kohnke T, Hoster E, Schneider S, Dufour A, Zellmeier E, Fiegl M, Braess J, Bohlander SK, Subklewe M, Sauerland MC, Berdel WE, Buchner T, Wormann B, Hiddemann W, Spiekermann K. Molecular response assessment by quantitative real-time polymerase chain reaction after induction therapy in NPM1-mutated patients identifies those at high risk of relapse. Haematologica. 2014 Aug;99(8):1317-25. doi: 10.3324/haematol.2014.104133. Epub 2014 May 9. PMID 24816240
- [Derived] Greif PA, Dufour A, Konstandin NP, Ksienzyk B, Zellmeier E, Tizazu B, Sturm J, Benthaus T, Herold T, Yaghmaie M, Dorge P, Hopfner KP, Hauser A, Graf A, Krebs S, Blum H, Kakadia PM, Schneider S, Hoster E, Schneider F, Stanulla M, Braess J, Sauerland MC, Berdel WE, Buchner T, Woermann BJ, Hiddemann W, Spiekermann K, Bohlander SK. GATA2 zinc finger 1 mutations associated with biallelic CEBPA mutations define a unique genetic entity of acute myeloid leukemia. Blood. 2012 Jul 12;120(2):395-403. doi: 10.1182/blood-2012-01-403220. Epub 2012 May 30. PMID 22649106